CLINICAL TRIAL: NCT02521389
Title: Assessment of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Oral Doses of Various Formulations of PWT-143 in Healthy Subjects
Brief Title: Assessment of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Various Formulations and Doses of PWT-143
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MEI Pharma, Inc. (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PWT-143
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Malignancies
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): 3 sequential groups (Groups A, B and C), comprising 3, 6 and 6 subjects, respectively, with 2 optional additional groups (Groups D and E), each comprising 6 subjects, to assess alternative dose levels or formulations (described below), if required.
  Interventions: Drug: PWT-143
- Part 2 (Experimental): Single dose, 2-way crossover design to assess a selected formulation of PWT-143 in the fed and fasted states in 8 subjects.
  Interventions: Drug: PWT-143

INTERVENTIONS:
Drug: PWT-143 — phosphatidylinositol-4,5-bisphosphate 3-kinase (PI3K) delta inhibitor

SUMMARY:
This single center first in human (FIH) study will comprise 2 parts; Part 1 will consist of 3 sequential dose groups (Groups A, B and C) and Part 2 will consist of 1 dose group (Group A). There will be an option to include 2 additional dose groups in Part 1 (Groups D and E) to assess alternative dose levels or formulations, if required.

In each study part, each subject will receive a single dose of investigational medicinal product PWT-143 in each of 2 study periods (total of 2 single doses).

DETAILED DESCRIPTION:
This first-in-human study will comprise 2 parts. In each part, each subject will receive a single dose of investigational medicinal product (IMP) in each of 2 study periods (total of 2 single doses).

Part 1 (Single Ascending Dose) This is an open-label, single dose design. It is planned to enroll up to 3 sequential groups (Groups A, B and C), comprising 3, 6 and 6 subjects, respectively, with 2 optional additional groups (Groups D and E), each comprising 6 subjects, to assess alternative dose levels or formulations (described below), if required.

The starting dose, dose increments and dose range are based on available pre-clinical data. Current planned dose levels are: 10, 30, 60, 90 and 150 mg (dose levels 1, 2, 3, 4 and 5, respectively); however, doses above 10 mg will be selected based on a review of emerging data from this study.

It is planned to use Formulation 1 for dose administration in Part 1 (Group A), selected from 3 test formulations. However, based on the exposure seen in the emerging data, an alternative formulation may be selected for dose comparison or escalation.

Part 2 (Food Effect Assessment) This is an open-label, randomised, single dose, 2-way crossover design to assess a selected formulation of PWT-143 in the fed and fasted states. Subjects will be administered a single dose of investigational medicinal product in the fed and fasted states across 2 study periods according to the randomisation schedule. There will be a minimum washout period for PWT-143 of 7 days between dose administrations in Periods 1 and 2.

It is planned that 1 group comprising 8 subjects will participate in Part 2. Subjects will be considered evaluable if they have received both treatments (ie, fed and fasted) and have completed safety assessments and PK sampling up to 24 h post-dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Age 18 to 65 years of age
3. Body mass index of 18.0 to 32.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
4. Part 2 only: Must be able to consume all food items in a standard high fat breakfast and/or have no conditions or surgery (eg, cholecystectomy) that could affect their ability to eat the high fat breakfast
5. Must be willing and able to communicate and participate in the whole study
6. Must be willing to provide voluntary written informed consent before performance of any study-related procedure that is not part of normal medical care
7. Must agree to use an adequate method of contraception

Exclusion Criteria:

1. Healthy males
2. Age 18 to 65 years of age
3. Body mass index of 18.0 to 32.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
4. Part 2 only: Must be able to consume all food items in a standard high fat breakfast and/or have no conditions or surgery (eg, cholecystectomy) that could affect their ability to eat the high fat breakfast
5. Must be willing and able to communicate and participate in the whole study
6. Must be willing to provide voluntary written informed consent before performance of any study-related procedure that is not part of normal medical care
7. Must agree to use an adequate method of contraception

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
The number of participants with and types of Adverse Events | 5 months

SECONDARY OUTCOMES:
Tmax (time from dosing at which Cmax is determined) | 5 months
Cmax (maximum observed plasma concentration) | 5 months
AUC (area under the concentration time curve) | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Pui Leung, MBChB, Principal Investigator — Study Principal Investigator
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom

REFERENCES:
- [Derived] Moreno O, Butler T, Zann V, Willson A, Leung P, Connor A. Safety, Pharmacokinetics, and Pharmacodynamics of ME-401, an Oral, Potent, and Selective Inhibitor of Phosphatidylinositol 3-Kinase P110delta, Following Single Ascending Dose Administration to Healthy Volunteers. Clin Ther. 2018 Nov;40(11):1855-1867. doi: 10.1016/j.clinthera.2018.09.006. Epub 2018 Oct 26. PMID 30458930